CLINICAL TRIAL: NCT00272376
Title: Clinical and Molecular Studies in Families With Myopia and Related Diseases
Brief Title: Clinical and Genetic Studies in Families With Myopia and Related Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060058; 06-EI-0058
Record Dates: First submitted 2006-01-05; First posted 2006-01-05 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2016-07-29

CONDITIONS: Myopia
Keywords: Myopia; Nearsightedness
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective

SUMMARY:
This study will examine the inheritance of myopia in families of various nationalities and ethnic backgrounds to identify gene changes that cause myopia or similar diseases and to better understand these conditions. In patients with myopia, the eye does not focus light accurately on the retina (tissue that lines the back of the eye), so that objects at a distance appear blurry. Myopia may occur alone, with other vision problems such as retinal dislocations, cataract or glaucoma, or with other problems such as joint or skin problems.

People with myopia (usually those from families with several affected members) and control subjects with normal vision may be eligible for this study.

Each participant undergoes the following procedures:

* Blood draw for genetic testing related to the disorders under study
* Medical and family history, including drawing a family tree to explore vision problems in the family
* Complete eye examination, including refraction (pupil dilation) and visual acuity testing, photographs of the retina and possibly lens, and specialized tests to measure field of vision, color vision and ability to see in the dark

DETAILED DESCRIPTION:
Objective: This project, Clinical and Molecular Studies in Families with Myopia and Related Diseases will study the inheritance of myopia in families of many nationalities and ethnic backgrounds in order to identify the genes that, when mutated, cause myopia, high myopia, or similar diseases and the pathophysiology through which they act.

Study Population: The number of subjects to be enrolled has no logical upper limit, but will be at least 250 and not more than 2000 during the next 5 years. The study consists of ascertaining individuals and especially families with multiple individuals, affected by myopia or related ocular diseases.

Design: These patients and their families will undergo detailed ophthalmological examinations and, where indicated, additional non-investigational examinations to characterize disease in their families and determine their affectation status. A blood sample will be collected from each individual for isolation of DNA and in some individual s biochemical studies or for lymphoblastoid transformation to establish a renewable source of DNA. Linkage analysis, physical mapping, and mutational screening will be carried out to identify the specific the gene and the mutations in it that are associated with myopia in this family. If necessary, the gene product or blood sample will be characterized biochemically. The study will enroll subjects at the NEI and at collaborating centers including the Zhongshan Ophthalmic Center of Sun Yat-Sen University, Guangzhou, China.

Outcome Measures: Linkage will be determined using the lod score method and mutations in specific genes will be assessed using a combination of residue conservation, blosum score, and molecular modeling. Biochemical, metabolic, and physiological effects will be individualized to the specific assay.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Individuals or family members of individuals with myopia, either congenital, childhood, or older.
  2. Adults must be capable of providing their own consent.
  3. All subjects must be able to cooperate with study examination and phlebotomy.
  4. Older than 4 years of age.

EXCLUSION CRITERIA:

1. Diseases, infections, or trauma that mimic primary myopia.
2. Children requiring sedation for study procedures.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2005-12-21; Study Completion 2016-07-29

PRIMARY OUTCOMES:
Statistically significant linkage

CONTACTS AND LOCATIONS:
Overall Officials: James F Hejtmancik, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzho, China

REFERENCES:
- [Background] Mutti DO, Mitchell GL, Moeschberger ML, Jones LA, Zadnik K. Parental myopia, near work, school achievement, and children's refractive error. Invest Ophthalmol Vis Sci. 2002 Dec;43(12):3633-40. PMID 12454029
- [Background] Teikari JM, O'Donnell J, Kaprio J, Koskenvuo M. Impact of heredity in myopia. Hum Hered. 1991;41(3):151-6. doi: 10.1159/000153994. PMID 1937488
- [Background] Zhang Q, Guo X, Xiao X, Yi J, Jia X, Hejtmancik JF. Clinical description and genome wide linkage study of Y-sutural cataract and myopia in a Chinese family. Mol Vis. 2004 Nov 17;10:890-900. PMID 15570218